CLINICAL TRIAL: NCT07061587
Title: Developing A Gout Action Plan in Primary Care Setting in Singapore
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Responsible Party: Principal Investigator, Liew Siew Lee, Family Physician, SingHealth Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0162
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Gout; Hyperuricemia; Gout Flare; Gout Chronic
Keywords: Gout action plan; action plan
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Intervention Model Description: The study will employ a sequential mixed-method design, which comprises of:
  1. Qualitative research to develop and refine prototype of gout action plan by gathering perspectives from both patients and healthcare providers.
  2. An open label pilot RCT to assess feasibility and estimate effectiveness of gout action plan in reducing gout flares, improvement in uric acid and quality of life.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Usual clinical care for this arm. No intervention delivered.
- Intervention arm (Active Comparator): Patients in intervention arm will receive gout action plan on top of usual clinical care.
  Interventions: Behavioral: Gout action plan

INTERVENTIONS:
Behavioral: Gout action plan — Gout action plan (that we aim to develop and refine during the study based on traffic light color system which will be categorized into zone system- green zone (well controlled), yellow zone (mild symptoms), red zone (severe symptoms). It will outline how to manage gout, identifying triggers, recognizing symptoms, appropriate medication usage, and when to seek medical attention)
  Arms: Intervention arm

SUMMARY:
The goal of this clinical trial is to develop a gout action plan in primary care setting in Singapore among adult patients with gout, and to learn if the gout action plan can improve gout control.

The main questions it aims to answer are:

* How do we develop a gout action plan in primary care setting in Singapore?
* What is the feasibility and estimate effectiveness of the developed gout action plan?
* Does gout action plan reduce frequency of gout flares in patients with gout?

Researchers will compare gout action plan to usual clinical care to see whether gout action plan helps in improving gout control.

Participants in intervention arm will be:

* given gout action plan and follow up for a course of 6 months
* asked to keep track of their gout symptoms
* follow up on the number of gout flares they have.

DETAILED DESCRIPTION:
Gout is a common inflammatory arthritis often seen in primary care. Worldwide prevalence ranges from under 1% to 6.8%.(1) The prevalence of gout has risen over the past three decades, accompanied by an increase in morbidity. (2) In Singapore, prevalence of gout is 4.1% amongst the Singapore Chinese population.(3) Gout is associated with significant morbidity and mortality due to coronary heart disease and kidney disease(3), and has substantial burden and impact in quality of life, with higher healthcare utilization and high unemployment rate observed in middle aged men with gout. (4)

Patients with poorly controlled gout suffer from frequent gout flares, with acute onset of joint pain and swelling, affecting health-related quality of life.(5) A meta-synthesis showed that gout flares impact on patients' lives, including physical, psychological, social and family life. (6) In a primary care institution in Singapore, 28.2% of patients with gout had poorly controlled disease.(7) In a rheumatology clinic in Singapore, 33% of patients with gout visited emergency department at least once for gout flare, while 19.5% had at least one hospitalization for gout.(4)

Acute gout flares can be mitigated by pharmacotherapy. Timely administration of acute medications is important to alleviate the pain leading to early resolution of symptoms. American College of Rheumatology (ACR) Guideline 2020 (8) and European League Against Rheumatism (EULAR) 2016 (9) recommend colchicine, non-steroidal anti-inflammatory drugs (NSAIDs) or corticosteroid for treatment of acute gout flare. In primary care clinics in Singapore, colchicine was often prescribed for an acute gout flare.(7) However, colchicine has gastrointestinal side effects such as vomiting and diarrhea (10), and some patients are not aware of its side effects and exceeded prescribed dose. (10) NSAIDs might improve the pain if given within 24 hours. (11) However, NSAIDs are associated with gastrointestinal, renal and cardiovascular adverse effects, thus they may not be the suitable pharmacotherapy for those with renal, gastrointestinal or cardiovascular comorbidities. (12) NSAIDs also cause hypersensitivity reactions with estimated prevalence of hypersensitivity to NSAIDs to be 0.5 to 1.9% of the general population. (13) For patients who are unable to tolerate NSAIDs or colchicine, or have chronic renal disease, systemic corticosteroid such as oral prednisolone might be a good alternative as it provides similar improvement in pain relief. (11,14)

Aside to pharmacotherapy, dietary control is important to prevent gout flares. ACG guideline 2020 (8) includes conditional recommendations to reduce alcohol intake, adopt a low-purine diet, and prioritize weight loss. A meta-analysis showed that red meat, seafood, alcohol, fructose or sweetened soft drinks increase risk of gout and hyperuricemia, while consumption of soy foods, dairy products and vegetables reduce risk of gout. (15) However, there is lack of awareness in dietary triggers especially in those with active gout. (16) A recent study in Australia found that patients with gout lack knowledge about the risk and protective factors of gout. (17) Patients resisted dietary changes due to the restrictive nature of the diet, lack of resources for information, and perceived it as unrealistic and unmanageable. (18 )

Gout control remains suboptimal despite established guideline. Urate lowering therapy (ULT) remains the key in gout management and its initiation is recommended for patients with recurrent gout flares with treat-to-target strategy. (8) However, in primary care institution in Singapore, it was found that half of the patients with poorly controlled gout were not prescribed urate lowering therapy.(7) In patients with gout, the overall adherence rate to ULT is as low as 47%.(19) Patients with gout demonstrate poor adherence to urate lowering therapy as they have limited knowledge of gout and its treatment, their attitude and perception towards taking long term medications. Some patients avoid ULT due to fear of side effects or flares during initiation, leading to nonadherence. (20)

Self-management is important in the management of chronic diseases. (21) Interventions of self-management have been shown to improve self-efficacy, health behavior, subsequently improving health status and quality of life and reducing healthcare utilization. (22) Self-efficacy refers to an individual's belief in their capacity to execute behaviors necessary to produce specific performance attainments, and it is correlated with self-care. Raising self-efficacy is important to change behavior in self-care. (23)

An action plan is a patient-held guide to support self-management with educational value. In chronic diseases such as asthma, the action plan provides information on how to manage the disease on a day-to-day basis and has proven to encourage self-management, improve health outcomes and quality of life, and reduce unscheduled visits to physicians. (24,25) Likewise, gout is a chronic condition with acute gout flares intermittently, that will benefit from self-management. In a study in Malaysia, patients were capable in self-management of gout but to variable extent, some practice diet control, some use painkillers during acute gout attacks, some use traditional medicine rather than taking allopurinol, some use exercise or stress-reducing activities, and the type of self-management might be influenced by cultural and social factors. (26)

To our knowledge, there is no well recognized gout action plan. A gout action plan has not been subjected to prior development in terms of content, design and acceptability. We hope that by developing a gout action plan, it will give information to patients about the disease to raise knowledge on gout, to reduce frequency of exacerbation via dietary control and lifestyle measures, to provide information on pain relief medications and the risks of taking painkiller, and urate lowering therapy for those with recurrent gout flares, and safety-netting advice on when to seek help. The study thus aims to develop a prototype of gout action plan by incorporating patients' and primary care physicians' perspectives, hoping to improve quality of life and healthcare utilization among patients with gout.

ELIGIBILITY:
For patient participants:

Inclusion Criteria:

* Adults who are 21 years old and above
* Clinical diagnosis of gout as per ACE-EULAR 2015 criteria
* Had at least an episode of gout exacerbation within the last 1 year
* Able to speak and read English
* Singapore citizens or permanent residents
* Able to provide informed consent

Exclusion Criteria:

* Mental disorders
* Cognitive impairment
* Hearing and/ or speech impairments
* Pregnant
* Known terminal illness
* Unable to provide informed consent

For healthcare professionals:

Inclusion Criteria (for healthcare professionals):

* Currently still in clinical practice
* Manage gout in their clinical practice

Exclusion Criteria (for healthcare professionals):

* Not involved in gout management in the practice
* No longer in clinical practice

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Creation of a gout action plan in primary care setting in Singapore | from enrolment to the end of in-depth interviews or focus group discussions at 6 months
  in-depth interviews or focus group discussions to develop and refine prototype of gout action plan by gathering perspectives from both patients and healthcare providers.

SECONDARY OUTCOMES:
Change from baseline in the number of gout flares at 6 months | from enrolment to the end of intervention at 6 months
  patient self-reported gout flares or visit to healthcare professionals for gout flares
Change of serum uric acid level from baseline at 6 months | from enrolment to end of intervention at 6 months
  serum uric level will be measured via laboratory test
change from baseline in health-related quality of life at 6 months | from enrolment to the end of intervention at 6 months
  participants achieved good quality of life on a scale ranging from 0 (worse quality of life) to 100 (best quality of life) using EQ-5D-5L questionnaire on health-related quality of life
Numbers of participants consented to join the study among those approached (participation rate) | from enrolment to end of intervention at 6 months
  participation rate will be counted at looking at proportion of participants consented to join the study compared to total number of participants approached to join the study
number of participants drop out of study (dropout rate) | from enrolment to end of intervention at 6 months
  dropout rate will be counted by looking at number of participants drop out of the study compared to number of participants consented

CONTACTS AND LOCATIONS:
Locations (1):
- SingHealth Polyclinics, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared as gout action plan is still yet to be developed and the study will firstly started with qualitative research to refine the prototype of gout action plan.

REFERENCES:
- [Result] Sivasegaran S, Hanafi NSH. Perceptions and practices of self-management among adult patients with gout at a primary care clinic: A qualitative study. Malays Fam Physician. 2023 Dec 18;18:72. doi: 10.51866/oa.428. eCollection 2023. PMID 38213387
- [Result] Hodkinson A, Bower P, Grigoroglou C, Zghebi SS, Pinnock H, Kontopantelis E, Panagioti M. Self-management interventions to reduce healthcare use and improve quality of life among patients with asthma: systematic review and network meta-analysis. BMJ. 2020 Aug 18;370:m2521. doi: 10.1136/bmj.m2521. PMID 32816816
- [Result] Gibson PG, Powell H, Coughlan J, Wilson AJ, Abramson M, Haywood P, Bauman A, Hensley MJ, Walters EH. Self-management education and regular practitioner review for adults with asthma. Cochrane Database Syst Rev. 2003;(1):CD001117. doi: 10.1002/14651858.CD001117. PMID 12535399
- [Result] Tan FCJH, Oka P, Dambha-Miller H, Tan NC. The association between self-efficacy and self-care in essential hypertension: a systematic review. BMC Fam Pract. 2021 Feb 22;22(1):44. doi: 10.1186/s12875-021-01391-2. PMID 33618661
- [Result] Allegrante JP, Wells MT, Peterson JC. Interventions to Support Behavioral Self-Management of Chronic Diseases. Annu Rev Public Health. 2019 Apr 1;40:127-146. doi: 10.1146/annurev-publhealth-040218-044008. Epub 2019 Jan 2. PMID 30601717
- [Result] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348
- [Result] Spragg JCJ, Michael TJF, Aslani P, Coleshill MJ, Chan JS, Day RO, Stocker SL. Optimizing adherence to allopurinol for gout: patients' perspectives. Br J Clin Pharmacol. 2023 Jul;89(7):1978-1991. doi: 10.1111/bcp.15657. Epub 2023 Jan 25. PMID 36607199
- [Result] Yin R, Li L, Zhang G, Cui Y, Zhang L, Zhang Q, Fu T, Cao H, Li L, Gu Z. Rate of adherence to urate-lowering therapy among patients with gout: a systematic review and meta-analysis. BMJ Open. 2018 Apr 10;8(4):e017542. doi: 10.1136/bmjopen-2017-017542. PMID 29643150
- [Result] Liddle J, Richardson JC, Hider SL, Mallen CD, Watson L, Chandratre P, Roddy E. 'It's just a great muddle when it comes to food': a qualitative exploration of patient decision-making around diet and gout. Rheumatol Adv Pract. 2021 Aug 13;5(3):rkab055. doi: 10.1093/rap/rkab055. eCollection 2021. PMID 34514294
- [Result] Chin A, Adams RJ, Gill TK, Hill CL. Gout Knowledge: A Survey of Australian Outpatients with Gout. Open Access Rheumatol. 2024 Jan 13;16:1-7. doi: 10.2147/OARRR.S435692. eCollection 2024. PMID 38239283
- [Result] Harrold LR, Mazor KM, Peterson D, Naz N, Firneno C, Yood RA. Patients' knowledge and beliefs concerning gout and its treatment: a population based study. BMC Musculoskelet Disord. 2012 Sep 21;13:180. doi: 10.1186/1471-2474-13-180. PMID 22995041
- [Result] Li R, Yu K, Li C. Dietary factors and risk of gout and hyperuricemia: a meta-analysis and systematic review. Asia Pac J Clin Nutr. 2018;27(6):1344-1356. doi: 10.6133/apjcn.201811_27(6).0022. PMID 30485934
- [Result] Rainer TH, Cheng CH, Janssens HJ, Man CY, Tam LS, Choi YF, Yau WH, Lee KH, Graham CA. Oral Prednisolone in the Treatment of Acute Gout: A Pragmatic, Multicenter, Double-Blind, Randomized Trial. Ann Intern Med. 2016 Apr 5;164(7):464-71. doi: 10.7326/M14-2070. Epub 2016 Feb 23. PMID 26903390
- [Result] Sanchez-Borges M, Caballero-Fonseca F, Capriles-Hulett A, Gonzalez-Aveledo L. Hypersensitivity Reactions to Nonsteroidal Anti-Inflammatory Drugs: An Update. Pharmaceuticals (Basel). 2010 Jan 5;3(1):10-18. doi: 10.3390/ph3010010. PMID 27713240
- [Result] Harirforoosh S, Asghar W, Jamali F. Adverse effects of nonsteroidal antiinflammatory drugs: an update of gastrointestinal, cardiovascular and renal complications. J Pharm Pharm Sci. 2013;16(5):821-47. doi: 10.18433/j3vw2f. PMID 24393558
- [Result] van Durme CM, Wechalekar MD, Landewe RB, Pardo Pardo J, Cyril S, van der Heijde D, Buchbinder R. Non-steroidal anti-inflammatory drugs for acute gout. Cochrane Database Syst Rev. 2021 Dec 9;12(12):CD010120. doi: 10.1002/14651858.CD010120.pub3. PMID 34882311
- [Result] Rebello C, Thomson M, Bassett-Clarke D, Martini N. Patient awareness, knowledge and use of colchicine: an exploratory qualitative study in the Counties Manukau region, Auckland, New Zealand. J Prim Health Care. 2016 Jun;8(2):140-8. doi: 10.1071/HC15023. PMID 27477556
- [Result] Richette P, Doherty M, Pascual E, Barskova V, Becce F, Castaneda-Sanabria J, Coyfish M, Guillo S, Jansen TL, Janssens H, Liote F, Mallen C, Nuki G, Perez-Ruiz F, Pimentao J, Punzi L, Pywell T, So A, Tausche AK, Uhlig T, Zavada J, Zhang W, Tubach F, Bardin T. 2016 updated EULAR evidence-based recommendations for the management of gout. Ann Rheum Dis. 2017 Jan;76(1):29-42. doi: 10.1136/annrheumdis-2016-209707. Epub 2016 Jul 25. PMID 27457514
- [Result] FitzGerald JD, Dalbeth N, Mikuls T, Brignardello-Petersen R, Guyatt G, Abeles AM, Gelber AC, Harrold LR, Khanna D, King C, Levy G, Libbey C, Mount D, Pillinger MH, Rosenthal A, Singh JA, Sims JE, Smith BJ, Wenger NS, Bae SS, Danve A, Khanna PP, Kim SC, Lenert A, Poon S, Qasim A, Sehra ST, Sharma TSK, Toprover M, Turgunbaev M, Zeng L, Zhang MA, Turner AS, Neogi T. 2020 American College of Rheumatology Guideline for the Management of Gout. Arthritis Care Res (Hoboken). 2020 Jun;72(6):744-760. doi: 10.1002/acr.24180. Epub 2020 May 11. PMID 32391934
- [Result] Oka P, Chong WM, Ng DX, Aau WK, Tan NC. Epidemiology and risk factors associated with gout control among adult Asians: a real-world retrospective cohort study. Front Med (Lausanne). 2023 Sep 7;10:1253839. doi: 10.3389/fmed.2023.1253839. eCollection 2023. PMID 37746085
- [Result] Stewart S, Guillen AG, Taylor WJ, Gaffo A, Slark J, Gott M, Dalbeth N. The experience of a gout flare: a meta-synthesis of qualitative studies. Semin Arthritis Rheum. 2020 Aug;50(4):805-811. doi: 10.1016/j.semarthrit.2020.06.001. Epub 2020 Jun 9. PMID 32554059
- [Result] Proudman C, Lester SE, Gonzalez-Chica DA, Gill TK, Dalbeth N, Hill CL. Gout, flares, and allopurinol use: a population-based study. Arthritis Res Ther. 2019 May 31;21(1):132. doi: 10.1186/s13075-019-1918-7. PMID 31151457
- [Result] Chua CKT, Cheung PP, Santosa A, Lim AYN, Teng GG. Burden and management of gout in a multi-ethnic Asian cohort. Rheumatol Int. 2020 Jul;40(7):1029-1035. doi: 10.1007/s00296-019-04475-6. Epub 2019 Nov 22. PMID 31758246
- [Result] Teng GG, Ang LW, Saag KG, Yu MC, Yuan JM, Koh WP. Mortality due to coronary heart disease and kidney disease among middle-aged and elderly men and women with gout in the Singapore Chinese Health Study. Ann Rheum Dis. 2012 Jun;71(6):924-8. doi: 10.1136/ard.2011.200523. Epub 2011 Dec 15. PMID 22172492
- [Result] He Q, Mok TN, Sin TH, Yin J, Li S, Yin Y, Ming WK, Feng B. Global, Regional, and National Prevalence of Gout From 1990 to 2019: Age-Period-Cohort Analysis With Future Burden Prediction. JMIR Public Health Surveill. 2023 Jun 7;9:e45943. doi: 10.2196/45943. PMID 37285198
- [Result] Dehlin M, Jacobsson L, Roddy E. Global epidemiology of gout: prevalence, incidence, treatment patterns and risk factors. Nat Rev Rheumatol. 2020 Jul;16(7):380-390. doi: 10.1038/s41584-020-0441-1. Epub 2020 Jun 15. PMID 32541923

DOCUMENTS (3):
  • Study Protocol (2025-03-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT07061587/Prot_000.pdf
  • Informed Consent Form: Patients (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT07061587/ICF_001.pdf
  • Informed Consent Form: Healthcare Professionals (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT07061587/ICF_002.pdf